CLINICAL TRIAL: NCT00369551
Title: A Safety and Feasibility Study of Bevacizumab With Paclitaxel, Carboplatin and Chest Radiotherapy in Patients With Locally Advanced Non-Small Lung Cancer
Brief Title: Bevacizumab, Paclitaxel, Carboplatin, and Radiation Therapy to the Chest in Treating Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02718; NCI-2012-02718 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-14576A; CDR0000491998; NCI-7213; 14576A (Other: University of Chicago); 7213 (Other: CTEP); P30CA014599 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Lung; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Stage II Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Paclitaxel; Taxes; Bevacizumab; Carboplatin

ARMS (1):
- Treatment (paclitaxel, carboplatin, bevacizumab, radiation) (Experimental): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, 36, and 43 and bevacizumab IV over 30-90 minutes on days 1, 15, 29, and 43. Patients also undergo chest radiotherapy 5 days a week for 7 weeks beginning on day 1.
  Consolidation therapy: Beginning 4-5 weeks after completion chemoradiotherapy, patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 1 hour followed by bevacizumab IV over 30 minutes. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Drug: paclitaxel; Biological: bevacizumab; Drug: carboplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies how well giving bevacizumab together with paclitaxel, carboplatin, and radiation therapy to the chest works in treating patients with locally advanced non-small cell lung cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab together with paclitaxel, carboplatin, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of administering bevacizumab, paclitaxel, carboplatin, and chest radiotherapy in patients with locally advanced non-small cell lung cancer.

II. Characterize the toxicity of this treatment regimen. III. Assess the clinical response to this treatment regimen. IV. Correlate circulating levels of angiopoietin-2 and vascular endothelial growth factor receptor-2 with clinical response to this treatment regimen.

OUTLINE: This is an open-label, multicenter study.Induction therapy.

Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, 36, and 43 and bevacizumab IV over 30-90 minutes on days 1, 15, 29, and 43. Patients also undergo chest radiotherapy 5 days a week for 7 weeks beginning on day 1.

Consolidation therapy: Beginning 4-5 weeks after completion chemoradiotherapy, patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 1 hour followed by bevacizumab IV over 30 minutes. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After study completion, patients are followed periodically for 36 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung carcinoma (NSCLC) meeting the following criteria:

  * The following subtypes are eligible:

    * Adenocarcinoma (including bronchoalveolar)
    * Large cell carcinoma (including giant and clear cell carcinomas)
    * Poorly differentiated carcinoma
  * No squamous cell histology
  * Unresectable stage II-III disease
  * Tumor must not invade the trachea or major arterial or venous structures
* Measurable or evaluable disease

  * Measurable disease defined as ? 1 lesion that can be accurately measured in ? 1 dimension as ? 20 mm with conventional techniques or as ? 10 mm with spiral CT scan
* No evidence of CNS disease, including primary brain tumor or brain metastases
* ECOG performance status (PS) 0-1 or Karnofsky PS 60-100%
* Life expectancy > 6 months
* Granulocyte count ? 1,500/mm³
* Platelet count ? 100,000/mm³
* Bilirubin < 1.25 times upper limit of normal (ULN)
* AST < 2.5 times ULN
* Creatinine normalOR creatinine clearance ? 60 mL/min
* FEV_1 ? 1.0 liters
* 24-hour urine protein < 1,000 mg (for patients with urine protein:creatinine ratio [by urine analysis] > 1.0)
* No hemoptysis within the past 12 months (defined as bright red blood in sputum of > 1 teaspoon)
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to carboplatin or taxane
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 14 days
* No clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident within the past 6 months
  * Uncontrolled hypertension
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Unstable angina pectoris
  * Clinically significant peripheral vascular disease
* No known bleeding diathesis or coagulopathy
* No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would limit study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ? 6 months after completion of study treatment
* No HIV positivity
* No prior chemotherapy
* No prior epidermal growth factor receptor-targeted therapy
* No prior vascular endothelial growth factor-targeted therapy
* No prior chest radiotherapy
* No major surgery or open biopsy within the past 14 days
* No concurrent treatment with full-dose anticoagulation

  * Low-dose anticoagulants (e.g., warfarin) to maintain patency of central venous catheter allowed provided all of the following criteria are met:

    * Daily dose of warfarin < 1 mg
    * INR < 1.5
* No other concurrent investigational agents
* No concurrent major surgical procedures
* No other concurrent anticancer agents or therapies
* No concurrent chronic treatment with aspirin (> 325 mg daily) or nonsteroidal anti-inflammatory agents
* No dexamethasone as an antiemetic during chemoradiotherapy
* No colony-stimulating factors during chemoradiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility | Up to 36 months
In-field toxicity, defined as bleeding or perforation of the tracheobronchial or gastrointestinal structures within the radiation field | Up to 36 months
Clinical response | Up to 36 months
Correlation of levels of angiopoietin-2 and vascular endothelial growth factor receptor-2 with clinical response | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States